CLINICAL TRIAL: NCT07297472
Title: Effect of Cold Application and Artificial Saliva in the Prevention of Chemotherapy-Induced Oral Mucositis in Patients With Cancer: A Randomized Controlled Trial
Brief Title: Effect of Cold Application and Artificial Saliva in the Prevention of Chemotherapy-Induced Oral Mucositis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karbala University (Other)
Responsible Party: Principal Investigator, Batool Abdulkareem Ahmed, Master's graduate student, Karbala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: prevention oral mucositis
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Oral Mucositis
Keywords: Cold application; Artificial saliva
MeSH Terms: conditions — Stomatitis | interventions — Cryotherapy; Saliva, Artificial

STUDY DESIGN:
Intervention Model Description: Cold application : Ice chips will be applied to the oral mucosa of the participants for 5 min before the chemotherapy session and 20 min during session than 5 min after the session.
  Artificial saliva: The patients will be asked to use the artificial saliva before breakfast, before lunch, before dinner and before bedtime. The patients will be given instructions on how to use the artificial saliva: they will be told to shake the bottle before use, to use enough artificial saliva to cover their whole mouth, to spray around their mouth, and to use their tongue to help spread the artificial saliva around their mouth.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cold application (Experimental): The participants asked to apply Ice chips to the oral mucosa for 5 min before the chemotherapy session and 20 min during session than 5 min after the session.
  Interventions: Other: cold application
- artificial saliva (Experimental): The participants asked to use the artificial saliva for 7 days before breakfast, before lunch, before dinner and before bedtime. The participants given instructions on how to use the artificial saliva: they told to shake the bottle before use, to use enough artificial saliva to cover their whole mouth, to spray around their mouth, and to use their tongue to help spread the artificial saliva around their mouth.
  Interventions: Other: Artificial Saliva
- control group (No Intervention): participants in the control group receive standard chemotherapy without cold application or artificial saliva

INTERVENTIONS:
Other: cold application — The participants asked to apply Ice chips to the oral mucosa for 5 min before the chemotherapy session and 20 min during session than 5 min after the session.
  Other Names: oral cryotherapy
  Arms: cold application
Other: Artificial Saliva — The participants asked to use the artificial saliva for 7 days before breakfast, before lunch, before dinner and before bedtime. The patients given instructions on how to use the artificial saliva: they told to shake the bottle before use, to use enough artificial saliva to cover their whole mouth, to spray around their mouth, and to use their tongue to help spread the artificial saliva around their mouth.
  Arms: artificial saliva

SUMMARY:
the Objectives of this clinical trial is :

1. To determine the effect of Cold Application for preventing of chemotherapy-Induced oral mucositis in cancer patients.
2. To examine the effect of artificial saliva for preventing of chemotherapy-Induced oral mucositis in cancer patients.
3. To compare between the effect of artificial saliva and cold application for preventing of chemotherapy-Induced oral mucositis in cancer patients.
4. To find out the differences between the effect of artificial saliva and cold application based on patient demographics and clinical data.

DETAILED DESCRIPTION:
The non-keratinized mucosa of the oral cavity including the tongue, buccal mucosa, and lips is particularly susceptible to injury, leading to ulcerative lesions clinically known as oral mucositis (OM). This common and impactful toxicity of standard cancer therapy, characterized by mucosal damage that can range from mild inflammation to deep ulceration.

In cases CIOM, the severity often requires major clinical interventions, including diet modification, opioid analgesics, and nutritional supplementation, to avoid disrupting optimal cancer therapy. Furthermore, CIOM can lead to superinfection, with the additional threat of bacteremia and sepsis. Patients with OM are more likely to experience negative treatment outcomes , and higher healthcare costs compared to those without the condition.

Oral mucositis (OM) notably reduces quality of life by causing both physical and psychological distress. This condition can lead to serious psychological issues like anxiety, depression, and social isolation. Moreover, pre-existing anxiety and depression may serve as risk factors for the development of oral mucositis. (Borowski et al., 2025).

Although the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO) have recommended some strategies, our knowledge regarding the prevention and treatment of CIOM remains limited, with no established evidence-based management regimens. This underscores the need to develop novel therapeutic drugs and strategies .

Cold application, commonly described as the cooling of the mouth during chemotherapy. is a valuable tool for preventing OM in patients receiving certain chemotherapeutic agents. It is safe and well-tolerated, and it can help to reduce the risk of complications .

Patients undergoing chemotherapy often develop transient or permanent xerostomia (subjective symptom of dry mouth) and hyposalivation (objective reduction of salivary flow). Hyposalivation can elevate tissue inflammation and thus increase the risk of local infection and make mastication difficult.as a result increased risk of developing severe OM .

Artificial saliva works by forming a continuous, proactive, and hydrating film that helps prevent OM .Most clinical studies of artificial saliva only focused on signs and symptoms of dry mouth . However, the effect of artificial saliva on oral mucositis has not directly established yet.

While both interventions show individual promise, it is reasonable that their mechanisms of action are complementary. Cold application preventing the initial cytotoxic effect and artificial saliva protecting and healing the compromised mucosa. However, there are lack of the sufficient evidence evaluating their combined effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo chemotherapy.
* Patients who do not have oral mucositis.
* Patients who are aged 18 years and older.
* Patients who are male or female.
* Patients who agree to be included in the study sample.

Exclusion Criteria:

* Patients who was refused to participate in the study.
* Patients who was not undergoing chemotherapy.
* Patients how was undergoing chemo-radiotherapy.
* Patients who selected for pilot study.

  * Patients diagnosed with oral mucositis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Challacombe Scale of Clinical Oral Dryness | Baseline and Day 7
  The Challacombe Scale is a clinician-administered tool for objectively assessing the severity of dry mouth (xerostomia) based on visual and tactile intraoral signs. It categorizes clinical oral dryness into ten grades (0 to 10), with increasing scores indicating greater severity. Key signs evaluated include mucosal appearance, saliva pooling, frothiness, and tongue features. This scale provides a standardized method to diagnose and monitor xerostomia
The World Health Organization (WHO) Oral Toxicity Scale | Baseline and Day 7
  The World Health Organization Oral Toxicity Scale, which was developed by the World Health Organization (WHO) in 1979. This scale categorizes oral mucositis (OM), a condition that involves inflammation and ulceration of the mucous membranes lining the oral cavity, into five different grades based on the severity of symptoms and their impact on diet and oral intake.
  Here is a brief overview of the five grades described in the scale. Grade 0: No Symptoms and diet is normal. Grade I: Soreness with or without erythematic (redness), and a solid diet is still possible.
  Grade II: Erythema and Ulcers present, and a soft or liquid diet is possible. Grade III: Confluent Ulcerations with or without exudates (discharge), and the person can only consume liquids.
  Grade IV: Deep Ulcerations and oral alimentation (consumption of food) is impossible. This grade is considered life-threatening.
Summated Xerostomia Inventory - SXI | Baseline and Day 7
  The Summated Xerostomia Inventory (SXI) is a validated patient-reported outcome measure (PROM) used to quantify the subjective symptoms of dry mouth (xerostomia).It composed of five items each item is scored on a five-point scale. Scoring is as follows: a Never response is scored as 1; Hardly ever scores 2; Occasionally scores 3; Frequently scores 4; and always scores 5. The scores for the 5 items are summed to give an overall SXI score which can range from 5 to 25. A higher score indicates more severe symptoms of xerostomia.

CONTACTS AND LOCATIONS:
Overall Officials: Batool A Ahmed, MSc, Principal Investigator — kerbala heath department

IPD SHARING:
Plan to Share IPD: No